CLINICAL TRIAL: NCT06597721
Title: First-in-Human, Phase 1 Study of ADCE-T02, a Tissue Factor Targeted Antibody-Drug Conjugate, in Patients With Advanced Solid Tumors
Brief Title: ADCE-T02, a Tissue Factor Targeted Antibody-Drug Conjugate, in Patients With Selected Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adcendo ApS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADCE-T02-001
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADCE-T02 Dose Escalation followed by an Expansion Phase (Experimental)
  Interventions: Drug: ADCE-T02

INTERVENTIONS:
Drug: ADCE-T02 — Administered intravenously

SUMMARY:
Adcendo ApS is conducting a phase 1 study of an investigational drug called ADCE-T02 (previously known as AMT-754), a tissue factor targeted antibody-drug conjugate which may be used in the future as a possible treatment for advanced solid tumors.

The main purpose of the study is to determine the Maximum Tolerated Dose (MTD), the recommended dose and the safety and tolerability of ADCE-T02 when given as a single therapy over a range of different dose levels.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients must have pathologically confirmed unresectable advanced solid tumor
2. Patients who have undergone at least one systemic therapy and have progressive disease
3. Patients must have at least one measurable lesion as per RECIST version 1.1.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
5. Life expectancy ≥ 3 months.
6. Patients must have adequate organ function as indicated by laboratory values
7. Women of childbearing potential (WCBP), defined as sexually mature women who have not undergone surgical sterilization or who have not been naturally postmenopausal for at least 12 consecutive months must agree to use two effective contraceptive methods while on study treatment and for at least 7 months after the last dose of ADCE T02.
8. Male patients must agree to use condoms, even if they have had a successful vasectomy, while on study treatment and for at least 4 months after the last dose of ADCE T02.

Key Exclusion Criteria:

1. Prior treatment with any agent targeting Tissue Factor or any ADC with a topoisomerase 1 payload
2. Central nervous system (CNS) metastasis.
3. Active ocular surface disease or a history of cicatricial conjunctivitis or inflammatory conditions that predispose to cicatrizing conjunctivitis, mucus pemphigoid or penetrating ocular transplants.
4. Persistent toxicities from previous systemic anti-neoplastic treatments
5. Known past or current coagulation defects leading to an increased risk of bleeding
6. Significant cardiac disease; recent myocardial infarction, acute coronary syndromes, congestive heart failure, uncontrolled hypertension, uncontrolled cardiac arrhythmias
7. History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, or current ILD/pneumonitis, or suspected ILD/pneumonitis
8. Prior second malignancy except for:

   * Well treated basal cell carcinoma or squamous cell carcinoma of the skin.
   * Low-risk prostate cancer with a Gleason score < 7 and a PSA level < 10 ng/mL
   * Any cancer or in situ cancer the patient has been disease-free for ≥ 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of ADCE-T02 | Up to 24 months
  The MTD will be determined using DLTs
Recommended Expansion Phase Dose (RED) of ADCE-T02 | Up to 24 months
  The RED will be determined using dose limiting toxicities (DLTs) and all other available study data
Type, incidence and severity of Adverse Events | Up to 24 months
  Safety and tolerability profile of ADCE-T02 assessed by the Common Terminology Criteria for Adverse Events v5.0

SECONDARY OUTCOMES:
Overall Response Rate (ORR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 24 months
  Proportion of patients achieving Complete Response (CR) or Partial Response (PR)
Disease Control Rate (DCR) according to the RECIST v1.1 | Up to 24 months
  Proportion of patients achieving CR, PR or Stable Disease (SD)
Progression-free Survival (PFS) | Up to 24 months
  Time from date of start of treatment to date of the first progression or death, whichever occurs first.
Concentration of anti-drug antibodies (ADA) | Up to 24 months
  Immunogenicity profile characterized by concentration of ADAs
Maximum observed concentration (C[max]) | Up to 24 months
  Pharmacokinetic profile characterized by the maximum observed concentration (C[max]) of ADCE-T02
Area under the curve (AUC) | Up to 24 months
  Pharmacokinetic profile characterized by the area under the curve (AUC) of ADCE-T02
Terminal half-life (t[1/2]) | Up to 24 months
  Pharmacokinetic profile characterized by the terminal half-life (t[1/2]) of ADCE-T02
Time to maximum concentration (Tmax) | Up to 24 months
  Pharmacokinetic profile characterized by the time to maximum concentration (Tmax)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (5):
  - Highlands Oncology Group, Rogers, Arkansas
  - Yale University Cancer Center, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas
  - START San Antonio, San Antonio, Texas
- Australia (5):
  - Scientia Clinical Research, Randwick, New South Wales
  - Southern Oncology Clinical Research Unit, Bedford Park, South Australia
  - Peninsula and South Eastern Haematology and Oncology Group (PSEHOG), Frankston, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Linear Clinical Research, Nedlands, Western Australia